CLINICAL TRIAL: NCT05767632
Title: An Open Label Randomized, Single Dose, Three-way, Partial Replicate Bioequivalence Study to Determine the Bioequivalence of Solifenacin Succinate & Mirabegron From Mirfenacin MR 5/50 mg Extended Release Tablets (Hikma Pharma, Egypt) Versus Vesicare 5 mg Film Coated Tablets & Betmiga 50 mg Prolonged-Release Tablets (Astellas Pharma Europe B.V, the Netherlands / Astellas Pharma Europe B.V, the Netherlands)
Brief Title: Bioequivalence Study of Solifenacin Succinate & Mirabegron From Mirfenacin MR 5/50 mg Extended Release Tablets (Hikma Pharma, Egypt) Versus Vesicare 5 mg FCT & Betmiga 50 mg Prolonged-Release Tablets (Astellas Pharma Europe B.V, the Netherlands / Astellas Pharma Europe B.V, the Netherlands)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: Hikma Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GRC/1/21/998
Record Dates: First submitted 2023-02-21; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — Solifenacin Succinate; mirabegron

STUDY DESIGN:
Intervention Model Description: An open label randomized, single dose, three-way, partial replicate crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- R reference (first dose) (Active Comparator): Reference drugs (Vesicare & Betmiga)
  Interventions: Drug: Vesicare (Solifenacin Succinate 5 mg) & Betmiga (Mirabegron 50 mg) (Reference first dose)
- T test (Experimental): Test drug (Mirfenacin MR)
  Interventions: Drug: Mirfenacin MR (Solifenacin Succinate 5 mg & Mirabegron 50 mg) (Test)
- R reference (second dose) (Active Comparator): Reference drugs (Vesicare & Betmiga)
  Interventions: Drug: Vesicare (Solifenacin Succinate 5 mg) & Betmiga (Mirabegron 50 mg) (Reference second dose)

INTERVENTIONS:
Drug: Vesicare (Solifenacin Succinate 5 mg) & Betmiga (Mirabegron 50 mg) (Reference first dose) — 1 tablet Vesicare contains Solifenacine succinate 5 mg & 1 tablet Betmiga contains Mirabegron 50 mg orally administrated followed by 240 ml of water
  Other Names: Vesicare & Betmiga
  Arms: R reference (first dose)
Drug: Mirfenacin MR (Solifenacin Succinate 5 mg & Mirabegron 50 mg) (Test) — 1 tablet Mirfenacin MR contains Solifenacine succinate 5 mg & Mirabegron 50 mg orally administrated followed by 240 ml of water
  Other Names: Mirfenacin MR
  Arms: T test
Drug: Vesicare (Solifenacin Succinate 5 mg) & Betmiga (Mirabegron 50 mg) (Reference second dose) — 1 tablet Vesicare contains Solifenacine succinate 5 mg & 1 tablet Betmiga contains Mirabegron 50 mg orally administrated followed by 240 ml of water
  Other Names: Vesicare & Betmiga
  Arms: R reference (second dose)

SUMMARY:
An open label randomized, single dose, three-way, partial replicate bioequivalence study to determine the bioequivalence of Solifenacin Succinate & Mirabegron From Mirfenacin MR 5/50 mg Extended Release Tablets (Hikma Pharma, Egypt) Versus Vesicare 5 mg Film Coated Tablets & Betmiga 50 mg Prolonged-Release Tablets (Astellas Pharma Europe B.V, the Netherlands / Astellas Pharma Europe B.V, the Netherlands)

DETAILED DESCRIPTION:
Healthy volunteers, 18-55 years of age, selected from the Egyptian population fulfilling the selection criteria. 30 Healthy volunteers (28 volunteers + 2 extra volunteers to compensate for drop-outs) will participate in the study. All dosed subject samples will be analyzed and their data will be included in the final study report.

For Solifenacin:

Primary Pharmacokinetic Parameters: Cmax and truncated AUC0→72 Secondary Pharmacokinetic Parameters: Tmax

For Mirabegron:

Primary Pharmacokinetic Parameters: Cmax, AUC0→t and AUC0→∞ Secondary Pharmacokinetic Parameters: Ke, tmax and t1/2e. ANOVA using 5% significance level for log transformed (with the 90% confidence intervals), untransformed data of Cmax, AUC0→t and AUC0→∞ and for untransformed data of Ke, tmax and t1/2e, for Mirabegron and untransformed data of Cmax and truncated AUC0→t and for untransformed data of tmax for Solifenacin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, age 18 to 55 years, inclusive.
2. Body weight within 15% of normal range (18.5-30.0) according to the accepted normal values for body mass index (BMI).
3. Medical demographics without evidence of clinically significant deviation from normal medical condition, eg.: no history of heart, liver, kidney, gastrointestinal, nervous system, or metabolic abnormalities.
4. Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
5. Females should be on a suitable birth control method.
6. Fully informed subjects that consented to participate in the study.

Exclusion Criteria:

1. Subjects with known allergy to the products tested.
2. Subjects who meet any of the contraindications to the administration of Solifenacin succinate and/or Mirabegron.
3. Subject does not agree not to consume any medication or food which may affect CYP3A4 enzyme at least two weeks prior to first study drug administration until donating the last sample of the study.
4. Subjects that do not agree not to consume alcohol-containing beverages and foods for 2 weeks before dosing and throughout the period of sample collection.
5. Heavy smokers.
6. Female subjects who were pregnant or nursing.
7. Acute infection within one week preceding first study drug administration.
8. History of drug or alcohol abuse.
9. Subject does not comply with the stated instruction of not taking any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
10. Subject is on a special diet (for example subject is vegetarian).
11. Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
12. Subject does not agree not to consume any beverages or foods containing grapefruit 14 days prior to first study drug administration until the end of the study.
13. Subject has a family history of severe diseases which have direct impact on the study.
14. Participation in a bioequivalence study or in a clinical study within the last 8 weeks before first study drug administration.
15. Subject intends to be hospitalized within 3 months after first study drug administration.
16. Subjects who have blood donated or lost more than 500 mL blood within 3 months prior to the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
For Solifenacin: Cmax | Up to 72 hours post dose in each treatment period
  to measure the maximal measured plasma concentration
For Solifenacin: truncated AUC0→72 | Up to 72 hours post dose in each treatment period
  to measure truncated area under the curve from zero time to 72 hours
For Mirabegron: Cmax | Up to 240 hours post dose in each treatment period
  to measure the maximal measured plasma concentration
For Mirabegron: AUC0→t | Up to 240 hours post dose in each treatment period
  to measure the area under the curve from zero time to 240 hours
For Mirabegron: AUC0→∞ | Up to 240 hours post dose in each treatment period
  to measure the area under the curve from zero time to infinity

SECONDARY OUTCOMES:
For Solifenacin & Mirabegron: Tmax | For Solifenacin:Up to 72 hours post dose in each treatment period & For Mirabegron:Up to 240 hours post dose in each treatment period
  Time of the maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshafeey, Ph.D. Pharma, Study Director — Genuine Research Center
Locations (1):
- Genuine Research Center GRC, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow SC, Wang H. On sample size calculation in bioequivalence trials. J Pharmacokinet Pharmacodyn. 2001 Apr;28(2):155-69. doi: 10.1023/a:1011503032353. PMID 11381568
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Background] Diletti E, Hauschke D, Steinijans VW. Sample size determination for bioequivalence assessment by means of confidence intervals. Int J Clin Pharmacol Ther Toxicol. 1991 Jan;29(1):1-8. PMID 2004861